CLINICAL TRIAL: NCT02365857
Title: Effects of Intrathecal Dexmedetomidine on the Perioperative Clinical Profile of Bupivacaine-induced Spinal Anesthesia for Cesarean Section
Brief Title: Intrathecal Dexmedetomidine With Bupivacaine for Spinal Anesthesia in Cesarean Section
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Professor Mohamed Abdulatif Mohamed, Abdulatif M., Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: thecaldex
Record Dates: First submitted 2015-02-04; First posted 2015-02-19 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2016-01

CONDITIONS: Anesthesia, Spinal
Keywords: spinal anesthesia; caesarian section; Dexmedetomidine
MeSH Terms: interventions — Dexmedetomidine; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- DEX-5 (Active Comparator): Dexmedetomidine & Bupivacaine. Patients will receive intrathecal 12.5 mg isobaric bupivacaine and 5 μg Dexmedetomidine using a total volume of injectate of 2.5 ml, and intrathecal injections will be given over approximately 10 to 15 seconds.
  Interventions: Drug: Dexmedetomidine & Bupivacaine.
- DEX-10 (Active Comparator): Dexmedetomidine & Bupivacaine. Patients will receive intrathecal 12.5 mg isobaric bupivacaine and 10 μg Dexmedetomidine using a total volume of injectate of 2.5 ml, and intrathecal injections will be given over approximately 10 to 15 seconds.
  Interventions: Drug: Dexmedetomidine & Bupivacaine.
- DEX-15 (Active Comparator): Dexmedetomidine & Bupivacaine. Patients will receive intrathecal 12.5 mg isobaric bupivacaine and 15 μg Dexmedetomidine using a total volume of injectate of 2.5 ml, and intrathecal injections will be given over approximately 10 to 15 seconds.
  Interventions: Drug: Dexmedetomidine & Bupivacaine.
- Control (Active Comparator): Bupivacaine Only. Patients will receive intrathecal 12.5 mg isobaric bupivacaine only using a total volume of injectate of 2.5 ml, and intrathecal injections will be given over approximately 10 to 15 seconds.
  Interventions: Drug: Bupivacaine Only.

INTERVENTIONS:
Drug: Dexmedetomidine & Bupivacaine. — Intrathecal injection of Dexmedetomidine & Bupivacaine.
  Arms: DEX-10; DEX-15; DEX-5
Drug: Bupivacaine Only. — Intrathecal injection of Bupivacaine only.
  Arms: Control

SUMMARY:
A Randomized, Controlled, Double blind study aiming to evaluate the analgesic potentials and side effect profile of different dose levels of Dexmedetomidine added to subarachnoid bupivacaine in full-term pregnant women undergoing elective cesarean section using spinal anesthesia. The investigators ultimate goal is to find out the least effective dose which will be associated with minimal or no side effects. The primary outcome will be the time to two sensory block segment regression.

DETAILED DESCRIPTION:
Alpha 2-agonists are non-opioid adjuvants with a significant role in extending the analgesic duration of subarachnoid block. When clonidine or Dexmedetomidine was added to intrathecal local anesthetics, the regression of sensory and motor blocks increased dose-dependently. Further, a recent meta-analysis including seven randomized controlled studies reported an increase in the duration of analgesia and reduced morphine requirement after the concomitant subarachnoid administration of clonidine.

Animal studies demonstrated that Dexmedetomidine added to bupivacaine significantly enhanced the duration of sensory and motor blockade of sciatic nerve block. Histo-pathological examination proved that all of the nerves analyzed had normal axons and myelin at 24 h and 14 days after the peri-neural administration of Dexmedetomidine. Several clinical studies confirmed the analgesic potentials and safe neurological outcome of neuraxially administered Dexmedetomidine in the non-obstetric settings while intrathecal clonidine proved to be a useful analgesic adjunct for spinal anesthesia in patients undergoing cesarean section. But to the best of the investigator knowledge the effects of intrathecal Dexmedetomidine on the perioperative clinical profile of bupivacaine-induced spinal anesthesia were not studied before in the obstetric patient population.

ELIGIBILITY:
Inclusion Criteria:

* Full-term pregnant women.
* Elective cesarean section using spinal anesthesia.
* Singleton gestation.
* American Society of Anesthesiologists (ASA) physical status classes I and II.

Exclusion Criteria:

* Preterm pregnancy (<37 wks gestation).
* Multiple gestation.
* Cardiovascular disease (e.g., preeclampsia, hypertension) and the use of antihypertensive medication.
* Conditions that preclude spinal anesthesia.
* Failed spinal block and conversion to general anesthesia.
* A history of established chronic pain.
* Drug addiction.
* A psychiatric disorder.
* Inability to communicate effectively.
* Asthma and allergy to non-steroidal anti-inflammatory drugs.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2014-12; Primary Completion 2015-07 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
The time to two sensory block segment regression. | 70 min
  Define the start of regression of the level of sensory block

SECONDARY OUTCOMES:
The peak sensory level of the block. | 10 min
  By Pin Prick testing.
Time from intrathecal injection to peak sensory block level. | 10 min
  Define the speed of onset of the block.
Time to S1 level sensory regression. | 70 min
  Define duration of the block.
Degree of motor block. | 24 h
  By Modified Bromage Score.
Intraoperative hemodynamic variables. | 24 h
  Detect frequency of side effects
The total dose of ephedrine/atropine required to maintain hemodynamic stability. | 24 h
  Detect frequency of side effects
The amount of lactated Ringer's solution required intraoperatively to maintain normal Blood pressure range | 24 h
  Detect frequency of side effects
Oxygen saturation (the need for O2 supplementation) | 24 h
  Detect frequency of side effects
Intraoperative analgesic supplementation | 70 min
  Define quality of the block
Time to first postoperative rescue analgesic request | 24 h
  Define duration of analgesia by the block
Postoperative pain scores for 24 hours | 24 h
  Define duration of analgesia by the block
Frequency of administration of postoperative analgesics | 24 h
  Define duration of analgesia by the block
Intraoperative sedation scores | 24 h
  Detect frequency of side effects
Incidence of side effects (nausea, vomiting, shivering, pruritus, respiratory depression, and desaturation) | 24 h
  Detect frequency of side effects
New born Apgar Score | 5 min
  Detect any effects on the new born at different dose levels
Duration of motor block. | 24 h
  By Modified Bromage Score.
Early postoperative hemodynamic variables. | 24 h
  Detect frequency of side effects
Total dose of postoperative analgesics | 24 h
  Define duration of analgesia by the block
Postoperative sedation scores | 24 h
  Detect frequency of side effects